CLINICAL TRIAL: NCT03875690
Title: Benefit of a Flash Dose of Corticosteroids in Digestive Surgical Oncology: a Randomized, Double Blind, Placebo-controlled Trial
Acronym: CORTIFRENCH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTEGA PHRCK 2017
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Elective Surgery for Any Digestive Cancer
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Injection of methylprednisolone; Biological: Blood samples
- Control group (Placebo Comparator)
  Interventions: Drug: Injection of sodium chloride; Biological: Blood samples

INTERVENTIONS:
Drug: Injection of methylprednisolone — Patients will receive 20mg/kg IV of methylprednisolone at the time of anaesthetic induction. Methylprednisolone will be infused in a ready-to-use 50 mL bag of sodium chloride 0.9% during 30 minutes at anaesthesic induction.
  Arms: Experimental group
Drug: Injection of sodium chloride — patients in the placebo group will receive 50 mL of sodium chloride 0.9% in a ready-to-use bag during 30 minutes at anaesthesic induction.
  Arms: Control group
Biological: Blood samples — electrolyte panel and glycemia performed within the first 24 hours after surgery.

SUMMARY:
Perioperative inflammation is harmful in cancer patients, namely in those undergoing surgery: it increases the risk of recurrence, decreases cancer survival, increases post-operative complications, and prolongs the time of recovery and the duration of hospital stay. Severe postoperative complications are also a risk factor of poor survival in cancer patients. Seemingly, some effective therapies currently used to improve the surgical outcome (e.g. immunonutrition, enhanced-recovery protocols) have an inflammatory effect. The modulation of perioperative inflammation therefore seems crucial to improve outcomes in patients undergoing surgery for digestive cancer.

A short perioperative treatment with high doses of corticosteroids has already been tested in several randomized trials. A recent meta-analysis showed that perioperative corticosteroids decreased inflammatory markers and might be associated with fewer complications in esophageal, liver, pancreatic and colorectal surgery: the decrease in the risk of postoperative complications was around 50% without adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age >_18 years
* Elective surgery for any digestive cancer (except purely hepatic surgery)
* Patients operated in a curative intent
* Patients who had given their written informed consent
* Patients affiliated to a National health insurance scheme

Exclusion Criteria:

* Emergency surgery
* Pregnant or breastfeeding women
* Patients with an ongoing oral treatment by steroids
* Palliative surgery
* Exclusive liver surgery
* Concomitant hyperthermic intraperitoneal chemotherapy
* Patient with at least one contra-indication to methylprednisolone treatment :
* active infection
* progressive/symptomatic viral infection (particularly hepatitis, herpes, chickenpox, herpes zoster)
* uncontrolled psychotic state
* hypersensitivity to methylprednisolone or to one of its excipients
* ASA grade >3
* Persons subject to a measure of legal protection (guardianship, tutorship)
* Persons subject to a court order
* Impossibility to adhere to the medical follow-up of the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
frequency of patients with postoperative major complications occurring within 30 days after surgery | Through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Dijon, Dijon, France

REFERENCES:
- [Derived] Magnin J, Fournel I, Doussot A, Regimbeau JM, Zerbib P, Piessen G, Beyer-Berjot L, Deguelte S, Lakkis Z, Schwarz L, Orry D, Ayav A, Muscari F, Mauvais F, Passot G, Trelles N, Venara A, Benoist S, Messager M, Fuks D, Borraccino B, Tresallet C, Valverde A, Souche FR, Herrero A, Gaujoux S, Lefevre J, Bourredjem A, Cransac A, Ortega-Deballon P. Benefit of a flash dose of corticosteroids in digestive surgical oncology: a multicenter, randomized, double blind, placebo-controlled trial (CORTIFRENCH). BMC Cancer. 2022 Aug 23;22(1):913. doi: 10.1186/s12885-022-09998-z. PMID 35999521